CLINICAL TRIAL: NCT03070275
Title: Preservation of Alveolar Crestal Bone From Implant Placement to Implant Exposure Using Autologous Alveolar Bone-Marrow Derived Mesenchymal Stem Cells (aBM-MSCs)
Brief Title: Dental Implant Placement in Adjunction With Autologous Alveolar Bone-Marrow Derived Mesenchymal Stem Cells (aBM-MSCs)
Acronym: Implant_bone
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Danae A. Apatzidou, Assist. Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ELKE_91480
Record Dates: First submitted 2017-02-25; First posted 2017-03-03 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Implant Therapy
Keywords: surgical implant placement; crestal bone; mucosa thickness; stem cells; fibrin glue; collagen fleece

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, single blind, control clinical trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor is not aware of the treatment modality
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group-A (Experimental): In the experimental Group (Group-A), a two-stage implant will be placed in parallel with an overlying biocomplex (aBM-MSCs/fibrin glue/collagen fleece) that comprises autologous alveolar bone marrow mesenchymal stem cells free of animal derived reagents, produced in clean room facilities and seeded into collagen scaffolds enriched with autologous fibrin glue.
  Interventions: Biological: Biocomplex: aBM-MSCs/fibrin glue/collagen fleece
- Control Group-B (Active Comparator): In Group-B, a two-stage surgical implant placement on the alveolar crest is followed based on the manufacturer's guidelines with no use of adjunctive grafting materials.
  Interventions: Procedure: Two-stage surgical implant placement

INTERVENTIONS:
Biological: Biocomplex: aBM-MSCs/fibrin glue/collagen fleece — Xeno-free, clinical-grade, autologous alveolar bone marrow mesenchymal stem cells enriched with autologous fibrin glue and loaded into a commercially available collagen fleece.
  Arms: Group-A
Procedure: Two-stage surgical implant placement — Implants are surgically placed on the alveolar crest following a two-stage protocol and the manufacture's guidelines with no adjunctives.
  Arms: Control Group-B

SUMMARY:
Systemically healthy volunteers with no active periodontal disease are recruited from referrals to the Dept. of Preventive Dentistry, Periodontology and Biology of Implants, Aristotle Univ of Thessaloniki for implant therapy. After signing a consent form, participants will be randomized into two treatment groups. Group-A (NA=10) will receive crestal placement of implants following a two-stage protocol in combination with a biocomplex comprising autologous alveolar bone marrow mesenchymal stem cells free of animal derived reagents, produced in clean room facilities and seeded into collagen scaffolds enriched with autologous fibrin glue. In Group-B (NB=10) implants are placed on the alveolar crest following a two-stage protocol and the manufacturer's guidelines. Intra-surgical clinical and radiographic assessments are performed at the time of implant placement (T0) and at the two-stage surgery (T1). Changes in mucosa thickness, width of keratinized tissues, marginal bone and bone thickness at the surgical site will be determined at T0-T1. Groups will be further divided into two subgroups based on mucosal thickness of the surgical site at T0 [thin mucosa (≤2.5mm) for Groups-AI/-BI; thick mucosa (>2.5mm) for Groups-AII/-BII]. A linear mixed model for repeated measures will be used for data analyses to determine changes in the dimensions of the peri-implant soft and hard tissues, around two stage-implants placed either conventionally, or in combination with the biocomplex.

DETAILED DESCRIPTION:
Aims & Objectives:

The present study describes a novel method to preserve the crestal bone at two-stage dental implants using autologous aBMMSCs, free of animal derived reagents, produced in clean room facilities enriched with autologous fibrin glue and seeded into commercially available collagen scaffolds (collagen fleece) that are stabilized over the implant platform upon surgical implant placement.

Primary objective:

This study aims to assess the efficacy of a novel method based on histotechnology in crestal bone preservation at two-stage dental implants, as compared to conventional surgical implant placement following the manufacturer's guidelines with no adjunctive use of grafting materials.

Secondary, changes in the peri-implant soft tissues will be also determined between implant placement and exposure and will be compared between the experimental and the conventional surgical treatment approaches.

Study design:

Biopsies will be derived from alveolar bone marrow of the alveolar bone under local anaesthesia in each patient belonging to the Experimental Group (Group-A). Briefly, after a thorough oral rinse with chlorhexidine 0.12% for 1min, an osteotomy using a trephine drill will be performed in the alveolar bone of an intraoral edentulous site other than the implant site and a 2x8 mm or 3cc approximately of an osseous core will be harvested. The area and the biopsy will be copiously irrigated with saline solution and then flaps will be sutured to achieve primary closure at the donor site. The bone sample will be then immediately placed in sterile tubes and will be transported to Biohellenika, Thessaloniki, Greece (http://www.biohellenika.gr) for stem cell isolation and expansion according to a strict clinical grade expansion protocol (Bakopoulou et al. 2013; Bakopoulou et al. in preparation). Since MSCs will be isolated and expanded in vitro in Good Laboratory Practice (GLP)-compliant clean rooms (Biohellenika facilities) meeting the quality guidelines set by the European Union and no animal derived reagents will be used throughout the experiments for autologous transplantation, the cells are considered safe for human clinical cell therapy applications. In Biohellenika facilities, 40ml of venous blood will be collected from each subject in Group-A shortly after the biopsy harvest, so that autologous serum is used for the isolation and culture expansion of the autologous stem cells. In addition, autologous fibrin glue will be used to load the BM-MSCs onto a commercially available collagen fleece. At the day of the surgical placement of the implants and chairside, the grafting material (BM-MSCs enriched with fibrin glue) will be delivered in an insulin syringe containing 10x10E6 cells/200μl fibrin and will be gently loaded onto the collagen fleece and activated with the addition of CaCl2. Subsequently, the biocomplex will be sutured onto the lingual flap using bioresorbable sutures (5-0 Coated VicrylTM (polyglactin 910), reverse cutting 3/8 circle - 16mm, Ethicon, Johnson & Johnson, New Brunswick, NJ, USA) and will be thus gently stabilized over the implant platform head partially covering the buccal bone. Handling of the scaffold will be done with care to avoid doing any harm to the viable cells.

In the Control Group (Group-B), the implants will be placed crestally following the manufacturer's guidelines with no adjunctive use of grafting materials. One system of implants will be consistently used throughout the study in both groups (Osseotite, Certain, parallel wall, Biomet 3i, Palm Beach Gardens, USA).

Post-operative care Post-operative pain will be controlled with Ibuprofen (600mg) at the end of the surgical procedure and 12h later if in pain. Amoxicillin (500mg / 8 hours for 5 days) will be prescribed to both Groups. All patients will be instructed to use 0.12% chlorhexidine twice daily and avoid brushing and chewing hard in the treated area for two weeks. During this 2-week period, patients will be followed on a weekly basis to record uneventful healing, and after that patients will discontinue rinsing with chlorhexidine solution and resume oral hygiene. Thereafter, subjects will be seen at three to four months to have their implants exposed.

Subjects will be assessed at baseline (T0: surgical implant placement) and T1 (implant exposure at 3-4 months). Clinical recordings will be determined by a single calibrated examiner using a manual periodontal probe (Hu-Friedy XP-23/QW, Hu-Friedy, Chicago, IL, USA) with an endo-stop attached on it and all measurements will be digitalised using an electronic caliper. A customised metallic caliper will measure the thickness of the bone at the buccal/lingual aspects of the implant. At T0 and T1, clinical recordings will assess:

1. Thickness of mucosa at the top of the alveolar ridge and 2- and 4mm apically, on the buccal and the lingual aspects of the ridge.
2. Width of keratinized mucosa buccally and lingually of the implantation site.
3. Thickness of buccal and lingual bone at 0, 3- and 6mm from the implant shoulder.
4. Level of of the buccal and lingual marginal bone, in relation to the implant shoulder.

Standardised digital radiographs will be collected at T0 and T1 to linearly determine changes (in mm) in the height of the alveolar bone between the implant shoulder and teh alveolar crest using the VixWin™ Platinum|Gendex software.

Groups will be further divided into two subgroups based on mucosal thickness of the surgical site at T0 [thin mucosa (≤2.5mm) for Groups-AI/-BI; thick mucosa (>2.5mm) for Groups-AII/-BII] and all the parameters will be determined and compared on the basis of the surgical approach and mucosa thickness at the surgical site.

A linear mixed model for repeated measures will be used for data analyses to determine changes in the dimensions of the peri-implant soft and hard tissues, around two stage-implants placed either conventionally, or in combination with the biocomplex.

ELIGIBILITY:
Inclusion Criteria:

• systemically healthy volunteers

Exclusion Criteria:

* poorly controlled systemic disease
* heavy smoking (>20cigs/day)
* bisphosphonate medication
* anti-inflammatory drugs
* bone metabolic diseases or disorders that compromise wound healing
* immunosuppressive therapy or radiation
* alcohol intake
* drug abuse over the past year
* significant concurrent illness
* pregnancy/lactation
* active periodontal disease and compromised oral hygiene (PI ≥25%)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
A reduction in the marginal bone levels | baseline (implant placement) to 4 months (implant exposure)
  Intra-surgical clinical data: Changes in the vertical distance from the implant shoulder to the alveolar crest in mm

SECONDARY OUTCOMES:
Radiographic changes in the marginal bone levels | baseline (implant placement) to 4 months (implant exposure)
  Radiographic data: linear measurements (mm) on standardised x-rays regarding vertical changes in the marginal bone levels from implant shoulder to the alveolar crest
Reduction in the thickness of the buccal/lingual bone | baseline (implant placement) to 4 months (implant exposure)
  Clinical data: Changes in the thickness of the bone plates in the buccal/lingual aspects of the implant
Changes in the alveolar mucosa | baseline (implant placement) to 4 months (implant exposure)
  Changes in the thickness of mucosa at the top of the alveolar ridge and at 2- and 4mm apically of the implant shoulder
Changes in the width of keratised mucosa | baseline (implant placement) to 4 months (implant exposure)
  Changes in the width of keratinised mucosa in mm at the surgical site

CONTACTS AND LOCATIONS:
Overall Officials: Antonis Konstantinidis, Professor, Study Chair — Retired, Dept. of Preventive Dentistry, Periodontology and Implant Biology, School of Dentistry, Aristotle University of Thessaloniki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakopoulou A, Leyhausen G, Volk J, Koidis P, Geurtsen W. Comparative characterization of STRO-1(neg)/CD146(pos) and STRO-1(pos)/CD146(pos) apical papilla stem cells enriched with flow cytometry. Arch Oral Biol. 2013 Oct;58(10):1556-68. doi: 10.1016/j.archoralbio.2013.06.018. Epub 2013 Jul 18. PMID 23871383